CLINICAL TRIAL: NCT00597246
Title: Imaging Brain Tumors With FACBC and Methionine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-028
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2019-06

CONDITIONS: Brain Cancer; CNS Cancer
Keywords: Brain; CNS; Central Nervous System
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Methionine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: FACBC, Methionine; Other: PET Scan

INTERVENTIONS:
Drug: FACBC, Methionine — F-18 labeled FACBC is prepared stereo-specifically in a semi-automated, NCA procedure utilizing the General Electric FDG MicroLab, a system employing a quaternary 4-aminopyridinium resin to effect F-18 fluorination. The triflate species is displaced with F-18 fluoride in the MicroLab, and then the 1-t-butyl carbamate-3- trifluoromethane sulfonoxy-1-cyclobutane-1-carboxylic acid methyl ester is hydrolyzed with 1 N HCl. The final product is isotonic and sterile, and has been utilized in animal experiments. The product was obtained in 30% radiochemical yield after 65 minutes from EOB. The radiochemical purity was greater than 95% and no preparative HPLC was required. The procedure could be considered routine, and is performed on the FDG synthetic module without changes either to the programming or to the cassettes.
Other: PET Scan — GE Advance PET scanner for sequential body imaging

SUMMARY:
This research protocol makes pictures of brain tumors. The pictures are made with a positron emission tomography (PET) scanner. PET scans use radioactivity to "see" cancer cells. We are using a new kind of PET scan. The new PET scan is called [18F]-FACBC PET. We will compare this to the standard PET scan. The standard PET scan is called [11C]-methionine PET.

We expect these pictures will give us information about your tumor. We also hope to collect information about the amount of radioactivity exposure. We will measure radioactivity exposure to your tumor, brain and other organs. The research study results will be used to support the submission of an investigational new drug (IND) application to the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The purpose of this research is to: 1) perform both 3-[18F]-FACBC and [11C-methyl]-Lmethionine brain tumor PET imaging studies in patients with primary brain tumors who have previously been treated and are now suspect for having recurrence or progression of disease (a pilot study, n=20); 2) perform only 3-[18F]-FACBC PET imaging studies on an additional set of patients with primary brain tumors who have previously been treated and are now suspect for having recurrence (n=10) . 3) obtain organ/tissue and body radiation dosimetry information following i.v. injection of 3-[18F]-FACBC; 4) look for potential correlations between the scan results obtained from those patients enrolled to 03-028 and the patients' past medical treatment; The first set of 20 patients will agree to two PET studies. One study will involve the i.v.

administration of a fluorine-18 labeled amino acid analogue, 3-fluoro-aminocyclobutane carboxylic acid (3-[18F]-FACBC) with sequential brain and body PET imaging. The second study will involve i.v. administration of [11C-methyl]-L-methionine and head imaging only.

The additional set of 10 patients will undergo one PET study which will consist of the i.v.

administration of fluorine-18 labeled amino acid analogue, 3-fluoro-aminocyclobutane carboxylic acid (3-[18F]-FACBC) with one brain scan and one body scan only. The 3-[18F]-FACBC PET studies (n=30) will be performed under the Radioactive Drug Research Committee (RDRC) guidelines as defined and established by the Federal Drug Administration (FDA). [11C-methyl]-L-methionine is in the hospital formulary and is approved for imaging brain tumors at MSKCC. Our hypotheses include: 1) [18F]-FACBC has equal or better brain tumor imaging characteristics compared to [11C]-methionine; 2) [18F]-FACBC is not metabolized, and radiolabeled metabolites will not confound the interpretation of the images as can be the case with [11C]-methionine; 3) imaging recurrent brain tumors with [18F]-FACBC will be enhanced by lower brain (background) activity as compared to corresponding [11C]- methionine images; 4) the biodistribution of [18F]-FACBC and radiation dosimetry following i.v. administration of a 370 MBq (10 mCi) dose is safe and within FDA guidelines; 5) a 370 MBq (10 mCi) dose of [18F]-FACBC is sufficient for imaging brain tumors in a clinical setting; 6) the accumulation of [18F]-FACBC will correlate with the patients response to prior treatment and will provide prognostic information with respect to tumor progression and survival.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient at MSKCC.
* Child-bearing age females must be non-pregnant, non-lactating, and must be using adequate contraception or surgically sterile.
* Karnofsky score of 60 or greater.
* Children that can sit still for 60-90 minutes, without sedation, will be included in this protocol.

Exclusion Criteria:

* Patient cannot tolerate lying still for 90 minute sessions in the PET tomograph.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-05-13 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald blasberg, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Brain Tumors: FACBC, Methionine: F-18 labeled FACBC is prepared stereo-specifically in a semi-automated, NCA procedure utilizing the General Electric FDG MicroLab, a system employing a quaternary 4-aminopyridinium resin to effect F-18 fluorination. The triflate species is displaced with F-18 fluoride in the MicroLab, and then the 1-t-butyl carbamate-3- trifluoromethane sulfonoxy-1-cyclobutane-1-carboxylic acid methyl ester is hydrolyzed with 1 N HCl. The final product is isotonic and sterile, and has been utilized in animal experiments. The product was obtained in 30% radiochemical yield after 65 minutes from EOB. The radiochemical purity was greater than 95% and no preparative HPLC was required. The procedure could be considered routine, and is performed on the FDG synthetic module without changes either to the programming or to the cassettes.
  PET Scan: GE Advance PET scanner for sequential body imaging
Period: Overall Study
Arm/Group | Participants With Brain Tumors
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Brain Tumors
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 54 [27 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Standardized Uptake Value of 3-[18F]-FACBC
Description: Determine clearance of 3-[18F]-FACBC in different tissues/organs of body.
Time Frame: Duration of scan, an average of 1 hour
Population: 3 participants did not receive 18F-Fluciclovine PET studies
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | Participants With Brain Tumors
Number analyzed (Participants) | 27
SUVmax | 4.5 (2.3)

2. Secondary Outcome: Rate of 18F-Fluciclovine Transport (k1) Into Tumors
Description: Look for potential correlations bet subsequent MR & PET results obtained from patients enrolled and patients' subsequent medical treatment, progression of tumor & survival.
Time Frame: Duration of scan, an average of 1 hour
Population: 3 participants did not receive PET scans
Measure: Mean (Standard Deviation); unit: mL/min/g
Arm/Group | Participants With Brain Tumors
Number analyzed (Participants) | 27
mL/min/g | 0.14 (0.24)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Participants With Brain Tumors
All-Cause Mortality (participants affected / at risk) | 29/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Brain Tumors (N=30)
Lymphopenia (Investigations) | 1
Prothrombin Time/PT (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT00597246/Prot_SAP_000.pdf